CLINICAL TRIAL: NCT05222698
Title: Segmental Free Latissimus Versus Free Gracillis Muscles Powered by Hypoglossal Nerve in Facial Reanimation of Long-standing Facial Palsy Patients
Brief Title: Free Neurovascularized Muscle Transfer in Facial Reanimation of Long-standing Facial Palsy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Saber Mahmoud, Assistant lecturer of plastic surgery, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-22-01-11
Record Dates: First submitted 2022-01-15; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Facial Paralysis
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Segmental free latissimus muscle trasfer to the face.
  Interventions: Procedure: Facial reanimation surgery by free muscle trasfer.
- Group B (Active Comparator): Free gracillis muscle trasfer to the face.
  Interventions: Procedure: Facial reanimation surgery by free muscle trasfer.

INTERVENTIONS:
Procedure: Facial reanimation surgery by free muscle trasfer. — Muscle flap harvesting from the back or from the thigh to be insetted to the paralyzed side of the face with microvascular anastomosis of the muscle pedicle to facial artery and vein.

SUMMARY:
The use of free Neurovascularized muscles like free latissimus and gracillis muscles for reanimation of long-standing facial palsy patients using the hypoglossal nerve for innervating these muscles

DETAILED DESCRIPTION:
The investigators need to know which of the two muscles is better functionally and aesthetically in facial reanimation of patients with facial paralysis of more than one year duration.

ELIGIBILITY:
Inclusion Criteria:

* All patients with facial paralysis more than one year what ever the cause.

Exclusion Criteria:

* patients with uncontrolled diabetes.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in smile excursion with the two muscles in the paralyzed side from the pre operative state. | One year post operatively.
  We will use SMILE system of Bray et al for assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Saber, Master, Principal Investigator — Sohag faculty of medicine

IPD SHARING:
Plan to Share IPD: No